CLINICAL TRIAL: NCT01618799
Title: An Open Label, Randomized, Two-Period, Two-Treatment, Two-Sequence, Crossover, Balanced, Single Dose Oral Bioequivalence Study of Lamotrigine Tablets 25 mg (2 × 25 mg Tablets) and 'LAMICTAL®' (Lamotrigine) Tablets 25 mg (2 × 25 mg Tablets) in Healthy Adult Human Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Lamotrigine Tablets 25 mg (2 x 25 mg Tablets) Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IPCA Laboratories Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Ipca/BA/1264033
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Fasting State
MeSH Terms: interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LAMICTAL® (Active Comparator): Lamictal® (Lamotrigine) Tablets 25 mg of GlaxoSmithkline, USA
  Interventions: Drug: Lamotrigine
- Lamotrigine Tablets 25 mg (Experimental): Lamotrigine Tablets 25 mg of M/s Ipca Laboratories Limited, India
  Interventions: Drug: Lamotrigine Tablets 25 mg

INTERVENTIONS:
Drug: Lamotrigine Tablets 25 mg — 2 x 25 mg tablet once a day
  Other Names: Test Product
  Arms: Lamotrigine Tablets 25 mg
Drug: Lamotrigine — 2 x 25 mg tablet once a day
  Other Names: LAMICTAL®
  Arms: LAMICTAL®

SUMMARY:
This is an open Label, randomized, two-period, two-treatment, two-sequence, crossover, balanced, single dose pivotal study. The purpose of this study is to assess the bioequivalence between Test Product and the corresponding Reference Product under fasting condition in healthy adult human subjects.

DETAILED DESCRIPTION:
Objective of this pivotal study was to assess the bioequivalence between Test Product: Lamotrigine Tablets 25 mg (2 x 25 mg)of M/s Ipca Laboratories Limited, India and the corresponding Reference Product: LAMICTAL® (Lamotrigine) Tablets 25 mg (2 x 25 mg) of GlaxoSmithkline, USA, under fasting condition in healthy adult human subjects in a randomized crossover study.

The study was conducted with 28 healthy adult subjects. In each study period, a single 2 X 25 mg dose of either test or reference was administered to the subjects as per the randomization schedule in each study period with about 240 mL of water at ambient temperature in sitting position.

The duration of the clinical phase was approximately 26 days including washout period of at least 21 days between administrations of study drug in each study period.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 45 years old, both inclusive.
2. Sex: Males and/or non-pregnant, non-lactating females.

   A. Females of childbearing potential must have a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test performed within 21 days prior to initiation of the study & prior to check-in of each period. They must be using an acceptable form of contraception.

   B. Acceptable forms of contraception include the following:

   i. Intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or

   ii. Barrier methods containing or used in conjunction with a spermicidal agent, or

   iii. Surgical sterilization or

   iv. Practicing sexual abstinence throughout the course of the study.

   C. Females will not be considered of childbearing potential if one one of the following is reported and documented on the medical history:

   i. Postmenopausal with spontaneous amenorrhea for at least one year, or

   ii. Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or

   iii. Total hysterectomy and an absence of bleeding for at least 3 months.
3. BMI: 18.5 to 24.9 weight in Kg / (height in meter)2 both inclusive; BMI value should be rounded off to one significant digit after decimal point (e.g. 24.94 rounds down to 24.9. while 18.45 rounds up to 18.5).
4. Able to communicate effectively with study personnel and willingness to follow the protocol requirements as evidenced by written informed consent.
5. Able to give written informed consent to participate in the study.
6. All volunteers must be judged by the principal or co-investigator or physician as normal and healthy during pre-study safety assessment performed within 21 days of the first dose of study medication which will include:

   1. A physical examination with no clinically significant finding.
   2. Results within normal limits or clinically non-significant for the tests mentioned in list of Laboratory Parameters:

      * Additional tests and/or examinations may be performed, if necessary, based on Principal Investigator discretion.
      * All results will be assessed against the laboratory normal ranges current at the time of testing and a copy of the normal ranges used will be included in the study documentation.

Exclusion Criteria:

1. History of allergic responses to Lamotrigine or other related drugs, or any of its formulation ingredients.
2. Have significant diseases or clinically significant abnormal findings during screening, [medical history, physical examination, laboratory evaluations, ECG, chest X-ray recording, obstetrics and gynecological history and examination along with PAP smear (for female volunteers) & transvaginal ultrasonography (for female volunteers)].
3. Any disease or condition which might compromise the haemopoeitic gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system, diabetes, psychosis or any other body system.
4. History or presence of bronchial asthma.
5. Use of any hormone replacement therapy within 3 months prior to study medication dosing.
6. A depot injection or implant of any drug within 3 months prior to administration of study medication.
7. Use of enzyme-modifying drugs within 30 days prior to receiving the first dose of study medication.
8. History or evidence of drug dependence or of alcoholism or of moderate alcohol use.
9. Smokers who smoke 10 or more cigarettes per day or 20 or more biddies per day or those who cannot refrain from smoking during the study period.
10. History of difficulty with donating blood or difficulty in accessibility of veins.
11. History of allergic response to heparin.
12. A positive hepatitis screen (includes subtypes B & C).
13. A positive test result for HIV antibody and / or syphilis (RPR/VDRL).
14. Volunteers who have donated blood (1 unit or 450 ml) within 90 days prior to the initial dose of the study drug or have blood loss, excluding volume drawn at screening for this study drug.
15. History of difficulty in swallowing, or of any gastrointestinal disease which could affect drug absorption.
16. Intolerance to venipuncture.
17. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Principal Investigator, could contraindicate the volunteer's participation in this study.
18. Volunteers who have received a known investigational drug within five elimination half life of the administered drug prior to the initial dose of study drug or who have participated in a clinical drug study or bioequivalence study within 90 days prior to initial dose of study drug, whichever is greater.
19. Found positive in urine test for drugs of abuse done before check-in of period I.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters. | 3 months
  Area Under Curve (AUC)and Cmax Sampling Hours: Pre-dose and at 00.25, 00.5, 00.75, 01.00, 01.25, 01.50, 01.75, 02.00, 02.25, 02.50, 03.00, 03.25, 03.50, 04.00, 04.25, 05.00, 06.00, 08.00, 10.00, 12.00, 18.00, 24.00, 36.00, 48.00 and 72.00 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Manish Singhal, MBBS, Principal Investigator — Cliantha Research Limited
Locations (1):
- Cliantha Research Limited, Ahmedabad, Gujarat, India